CLINICAL TRIAL: NCT06296810
Title: Implementation of Adaptive DBS to Offset STN Dysregulation During Exercise and Reduce Exertion in Parkinson's Disease
Brief Title: Adaptive DBS to Offset STN Dysregulation During Exercise in PD
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0847
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- PD: Subjects with PD who have an implanted Medtronic DBS system with a Percept IPG.
  Interventions: Device: aDBS

INTERVENTIONS:
Device: aDBS — adaptive deep brain stimulation

SUMMARY:
The investigators conduct a prospective study to evaluate the effects of exercise on Parkinson's Disease brain biomarkers detected with the PerceptTM PC neurostimulator.

DETAILED DESCRIPTION:
The investigators will conduct a prospective study to evaluate the effects of exercise on Local Field Potential biomarkers detected from the subthalmic nuclues in Parkinson's Disease with the PerceptTM PC neurostimulator. Subsequently, adaptive Deep Brain Stimulation applied in response to low beta peak (L-beta; 13-20Hz) will be performed to evaluate feasibility of whether aDBS can offset the effects of exacerbation of parkinsonism during exercise performance and recovery.

ELIGIBILITY:
Inclusion Criteria:

Persons with PD who have a Medtronic DBS Sensight implant and a Percept IPG.

-

Exclusion Criteria:

Persons not meeting the above listed implant criteria Persons not meeting the age limit criteria Persons who are not able to complete the study exercise Persons not able to comprehend and consent to study participation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with PD, who have a Medtronic DBS Sendight implant and a Percept IPG.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
identification of L-beta frequency peak power | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Aurora, Colorado, United States